CLINICAL TRIAL: NCT00356408
Title: An Open-label, Multi-center Trial to Examine the Long Term Safety, Efficacy, and Corticosteroid-sparing Effect of Certolizumab Pegol in Patients With Moderate to Severe Crohn's Disease Previously Enrolled in C87059 (COSPAR I, NCT00349752).
Brief Title: Examining the Long Term Safety, Efficacy, and Corticosteroid-sparing Effect of Certolizumab Pegol in Crohn's Disease
Acronym: COSPAR II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87065; 2006-003871-11 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2011-04

CONDITIONS: Crohn's Disease
Keywords: CDP870; certolizumab pegol; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDP870 400 mg (Experimental): Certolizumab pegol (CDP870) 400 mg (2 injections of 1 mL) every 4 weeks from Week 2 until Week 34, or until CDP870 is available for a Crohn's disease indication in the patient's country. Subjects who were Non-completers of C87059 (COSPAR I, NCT00349752) receive an additional CDP870 400 mg dose at Week 2
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — Certolizumab pegol (CDP870), an anti-tumor necrosis factor (TNF)α, humanized antibody Fab' fragment - polyethylene glycol conjugate, solution for injection, in 10 mM sodium acetate buffer and 125 mM sodium chloride, pH 4.7, supplied in 3 mL vials with a fill of 1.4 mL (an extractable volume of 1 mL corresponds to a dose of 200 mg).
  Dosing is every 4 weeks from Week 2 until Week 34, or until CDP870 is available for a Crohn's disease indication in the patient's country. Subjects who were Non-completers of C87059 (COSPAR I, NCT00349752) receive an additional CDP870 400 mg dose at Week 2.
  Other Names: CDP870; CZP; Cimzia

SUMMARY:
This is an open-label extension study designed to measure the safety, efficacy, and corticosteroid-sparing effect of certolizumab pegol (CDP870) in patients with moderate to severe Crohn's disease previously enrolled in C87059 (COSPAR I, NCT00349752).

ELIGIBILITY:
Inclusion Criteria:

* Patients previously enrolled in C87059 (COSPAR I, NCT00349752)

Exclusion Criteria:

* Subject withdrawn or discontinued from C87059 (COSPAR I, NCT00349752) study under specific conditions
* Subject who received treatment other than study medication and other than medications permitted in C87059 (COSPAR I, NCT00349752)
* Subjects from countries where certolizumab pegol is authorized in Crohn's disease treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (63):
- United States (49):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - La Jolla, California
  - Oceanside, California
  - Palo Alto, California
  - Roseville, California
  - Lakewood, Colorado
  - Clearwater, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - North Miami Beach, Florida
  - Marietta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Bloomington, Indiana
  - Davenport, Iowa
  - Topeka, Kansas
  - Bowling Green, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Annapolis, Maryland
  - Newton, Massachusetts
  - Chesterfield, Michigan
  - Dearborn, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Kansas City, Missouri
  - Mexico, Missouri
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Austin, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin
- Canada (9):
  - Edmonton, Alberta
  - Abbottsford, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
  - Calgary
- Germany (5):
  - Frankfurt
  - Heidelberg
  - Jena
  - Rostock
  - Ulm

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was started in January 2007 with recruitment occurring in the United States, Germany, and Canada. The study had last patient last visit in February of 2010.
Period: Overall Study
Arm/Group | CDP870 400 mg
Started | 103 (106 subjects enrolled, however only 103 were included in the Intent to Treat (ITT) population.)
Completed | 43
Not Completed | 60
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 36
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6
Not completed — Other: Principal investigator discretion | 3
Not completed — Other: Sponsor request | 1
Not completed — Other: Azathioprine stopped | 1
Not completed — Other: Failed to meet Inc/Exc criteria | 1
Not completed — Other: Subject chose commerical dosing | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Completer: Placebo Completer: Placebo subjects who completed C87059. Regardless of their remission status and steroids use, they have participated to the week 38 visit of C87059.
- CDP870/Completer: CDP870 Completer: CDP870 subjects who completed C87059. Regardless of their remission status and steroids use, they have participated to the week 38 visit of C87059.
- Placebo/Non-completer: Placebo Non-completer: Placebo subjects who left C87059 early because of failure (relapse/treatment failure or not tolerating the Corticosteroids tapering/needing reintroduction of Corticosteroids).
- CDP870/Non-completer: CDP870 Non-completer: CDP870 subjects who left C87059 early because of failure (relapse/treatment failure or not tolerating the Corticosteroids tapering/needing reintroduction of Corticosteroids).
- Total: Total of all reporting groups
Arm/Group | Placebo/Completer | CDP870/Completer | Placebo/Non-completer | CDP870/Non-completer | Total
Number analyzed (Participants) | 14 | 16 | 40 | 33 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 39 | 32 | 101
  >=65 years | 0 | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.00 (12.53) | 39.31 (12.83) | 38.44 (13.73) | 41.38 (13.75) | 40.27 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 22 | 18 | 55
  Male | 8 | 7 | 18 | 15 | 48
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 31 | 21 | 70
  Canada | 4 | 6 | 7 | 10 | 27
  Germany | 2 | 0 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of at Least One Treatment-emergent Adverse Event During This Study (Maximum 122 Weeks)
Description: Results are presented as the number of subjects with at least one treatment-emergent adverse event during this study.
Time Frame: During this study (maximum 122 weeks)
Population: All subjects in the the Intent to Treat (ITT) population are included in this analysis.
Measure: Number; unit: subjects
Arm/Group | Placebo/Completer | CDP870/Completer | Placebo/Non-completer | CDP870/Non-completer
Number analyzed (Participants) | 14 | 16 | 40 | 33
subjects | 12 | 15 | 32 | 30

2. Secondary Outcome: Disease Remission (Crohn's Disease Activity Index, CDAI≤150) at Week 34 in Patients Who Completed/Did Not Complete C87059 (COSPAR I, NCT00349752) and Remained Off Corticosteroids.
Description: Crohn's disease activity index (CDAI) is used to quantify the symptoms of Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease. Results are presented as the percentage of subjects in disease remission at Week 34.
Time Frame: Week 34 in this study
Population: All subjects in the the Intent to Treat (ITT) population are included in this analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo/Completer | CDP870/Completer | Placebo/Non-completer | CDP870/Non-completer
Number analyzed (Participants) | 14 | 16 | 40 | 33
percentage of subjects | 28.6 | 37.5 | 35.0 | 3.0

ADVERSE EVENTS:
Time Frame: Duration of the study, maximum of 122 Weeks
Groups:
- Placebo/Completer: Placebo Completer: Placebo subjects who completed C87059. Whatever their remission status and steroids use, they have participated to the week 38 visit of C87059.
- CDP870/Completer: CDP870 Completer: CDP870 subjects who completed C87059. Whatever their remission status and steroids use, they have participated to the week 38 visit of C87059.
- CDP870 400 mg (Overall): Certolizumab pegol (CDP870) 400 mg (2 injections of 1 mL) every 4 weeks from Week 2 until Week 34, or until CDP870 is available for a Crohn's disease indication in the patient's country. Subjects who were Non-completers of C87059 (COSPAR I, NCT00349752) receive an additional CDP870 400 mg dose at Week 2
Arm/Group | Placebo/Completer | CDP870/Completer | Placebo/Non-completer | CDP870/Non-completer | CDP870 400 mg (Overall)
Serious Adverse Events (participants affected / at risk) | 5/14 | 0/16 | 6/40 | 4/33 | 15/103
Other Adverse Events (participants affected / at risk) | 11/14 | 15/16 | 31/40 | 27/33 | 84/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Completer (N=14) | CDP870/Completer (N=16) | Placebo/Non-completer (N=40) | CDP870/Non-completer (N=33) | CDP870 400 mg (Overall) (N=103)
Crohn's Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (6) | 1 (1) | 5 (8)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Perianal Abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Completer (N=14) | CDP870/Completer (N=16) | Placebo/Non-completer (N=40) | CDP870/Non-completer (N=33) | CDP870 400 mg (Overall) (N=103)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Cerumen Impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 8 (11) | 11 (13) | 22 (27)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 6 (6) | 11 (11)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (2) | 3 (4) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (11) | 2 (3) | 7 (16)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (6)
Rectal Haemorrhage (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (3) | 0 (0) | 6 (8)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 5 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (4)
Tooth Impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (4)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dental Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (3) | 8 (9)
Fatigue (General disorders) | 1 (3) | 1 (1) | 2 (2) | 2 (2) | 6 (8)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Influenza Like Illness (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Injection Site Pain (General disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 3 (5)
Injection Site Irritation (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Injection Site Erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 6 (7) | 5 (7) | 14 (17)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 7 (9) | 3 (4) | 12 (15)
Sinusitis (Infections and infestations) | 1 (1) | 3 (4) | 5 (6) | 1 (1) | 10 (12)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (5) | 8 (9)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 4 (7) | 1 (1) | 7 (10)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (4)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Exposure To Toxic Agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Blood Creatinine Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzyme Abnormal (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6) | 8 (11) | 7 (8) | 19 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 7 (8)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 5 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 3 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 5 (7) | 5 (6) | 11 (14)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 7 (7)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (12) | 6 (17)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 6 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Stress (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (2) | 3 (4) | 6 (9)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vascular Skin Disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.